CLINICAL TRIAL: NCT06405594
Title: Neurocognitive Mechanisms of Sentence Production Impairment in Aphasia
Acronym: sentence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Yasmeen Faroqi Shah, Professor, University of Maryland, College Park
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2044118-1
Record Dates: First submitted 2024-05-01; First posted 2024-05-08 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Aphasia, Acquired; Stroke; Healthy Aging
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Intervention Model Description: All participants will receive the same intervention (language condition) and a single arm (language condition)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Language condition (Experimental): All participants will receive this arm. In this arm, the intervention involves asking participants to speak and understand words and sentences with different linguistic manipulations such as morphological, semantic, phonological priming, predictability of the subject and object nouns associated with verbs, naming of verbs and nouns, production of sentences with past, future or present tense. Accuracy, response times and brain activity are the outcome measures.
  Interventions: Behavioral: Language Condition

INTERVENTIONS:
Behavioral: Language Condition — The intervention involves asking participants to speak and understand words and sentences with different linguistic manipulations such as morphological, semantic, phonological priming, predictability of the subject and object nouns associated with verbs, naming of verbs and nouns, production of sentences with past, future or present tense. Accuracy, response times and brain activity are the outcome measures.

SUMMARY:
The proposed research is relevant to public health because stroke is a leading cause of long-term disability among older adults and communication impairments resulting from stroke have a significant negative impact on quality of life. By seeking to better understand post-stroke aphasia, this project lays the groundwork for development of new interventions, and aligns with NIDCD's priority areas 1 (understanding normal function), 2 (understanding diseases), and 3 (improving diagnosis, treatment, and prevention).

DETAILED DESCRIPTION:
Post-stroke agrammatic aphasia (PSA-G) is characterized by a cluster of symptoms (fragmented sentences, errors in functional morphology, a dearth of verbs, and slow speech rate), yet extant theories and language interventions focus on individual symptoms. This single-symptom theoretical and intervention focus results in limited gains in functional communication. The long-term goal of this research is to improve the clinical effectiveness of interventions for PSA-G.

As a first step towards this goal, this project's objective is to advance the theoretical framework of PSA-G by addressing two critical gaps. The first gap is in the mechanistic understanding of how lexical, grammatical, motoric, and cognitive processes work together to enable fluent sentence production and how this breaks down in PSA-G. The second gap is in the understanding of neural mechanisms underlying how sentence production planning normally unfolds over time and what crucial spatiotemporal alterations give rise to PSA-G versus other variants of post-stroke aphasia with predominantly lexico-semantic deficits (PSA-LS). The central hypothesis is that agrammatic language production results from spatiotemporal alterations in the neural dynamics of morphosyntactic and phonomotor processes, causing a cumulative processing bottleneck at the point of articulatory planning. This Synergistic Processing Bottleneck Model of Agrammatism will be tested with two specific aims.

Specific Aim 1 will elucidate the relative contribution of syntactic and non-syntactic processes towards sentence production in aphasia by using speed metrics and a path modeling framework. The expected outcomes of this aim are an improved understanding of the extent to which delays in different linguistic processes underlying the agrammatic symptom cluster impair fluent sentence production in aphasia generally, and in PSA-G versus PSA-LS more specifically.

Specific Aim 2 will determine the neural mechanisms underlying sentence production across language deficit profiles. Magnetoencephalography (MEG) will be used to compare alterations in timecourse and functional connectivity of key perilesional and contralesional syntactic hubs across increasingly demanding morphosyntactic production tasks. The expected outcome of this aim is a spatiotemporally specified neural model of sentence production in neurotypical, PSA-G, and PSA-LS speakers.

The significance this research is that it will forward an empirically established multidimensional model of sentence production, which will lay the foundation for developing more targeted and effective language interventions for agrammatic aphasia. It will also contribute to a better understanding of agrammatism in neurodegenerative aphasias. The innovative aspects of this project include: a novel multidimensional theoretical framework that incorporates non-syntactic dimensions of phonomotor planning, processing capacity and speed, and neurophysiological dynamics; direct comparisons between PSA-G and PSA-LS groups; and MEG analysis of spoken language with simultaneous electromyographic measurement.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Persons with acquired aphasia are defined as those with a language impairment following left hemisphere brain injury (most likely a stroke).
* Neurotypical adults need to be either young (ages 18-30 years) or older (> 60 years)
* Native (or primary) speakers of English

Exclusion Criteria:

* Prior neurological or psychiatric diagnoses or developmental disabilities before the onset of aphasia
* do not speak English fluently

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Accuracy | through the completion of the study, an average of 1 year
  Response accuracy for each experimental condition will be measured
Response time | through the completion of the study, an average of 1 year
  Response times for each experimental condition will be measured
Brain activity | through the completion of the study, an average of 1 year
  Patterns of brain activity (using magnetoencephalography and MRI) will be measured for each experimental condition

CONTACTS AND LOCATIONS:
Overall Officials: Yasmeen Faroqi-Shah, PhD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, College Park, Maryland, United States